CLINICAL TRIAL: NCT06862960
Title: Ozanimod for the Treatment of Alzheimer's Disease: a Proof-of-concept Study
Brief Title: Ozanimod in Patients With Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ChenXiaoChun (Other)
Collaborators: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor-Investigator, ChenXiaoChun, Professor, Fujian Medical University Union Hospital
Organization: Fujian Medical University Union Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024XHYG0025
Record Dates: First submitted 2025-03-05; First posted 2025-03-07 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Ozanimod; sphingosine-1-phosphate receptor; cognitive dysfunction
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ozanimod Group (Experimental): Patients will receive ongoing approved AD treatment (eg, acetylcholinesterase inhibitors, memantine, or both) plus ozanimod. Ozanimod will be administered in strict accordance with the stepwise dose-escalation protocol (Days 1-4: 0.23 mg/day; Days 5-7: 0.46 mg/day), followed by a maintenance dose of 0.92 mg once daily from Day 8. The total treatment duration will be 27 weeks, including both titration and maintenance phases.
  Interventions: Drug: Ozanimod
- Control Group (Active Comparator): Patients will receive ongoing approved AD treatment (eg, acetylcholinesterase inhibitors, memantine, or both).
  Interventions: Drug: Conventional medication

INTERVENTIONS:
Drug: Ozanimod — A sphingosine-1-phosphate receptor regulator
  Arms: Ozanimod Group
Drug: Conventional medication — Conventional medications for moderate AD
  Arms: Control Group

SUMMARY:
The purpose of this study is to investigate the benefits of ozanimod in patients with moderate Alzheimer's disease.

DETAILED DESCRIPTION:
This study will enroll 40 patients with moderate Alzheimer's disease (AD), who will be divided into two groups according to a fixed 1:1 (ozanimod : control) schedule. Patients in control group will receive ongoing approved AD treatment (eg, acetylcholinesterase inhibitors, memantine, or both), while those in the ozanimod group will receive the same approved AD treatment with the addition of ozanimod. The treatment will be for 27 weeks. All participants will undergo assessments at baseline and week 27, including 18F-florbetaben PET imaging, blood tests, and cognitive evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Must meet the 2024 diagnostic criteria for Alzheimer's disease (AD) published by the Alzheimer's Association (AA), and be in the moderate stage of AD.
2. The Clinical Dementia Rating-Sum of Boxes (CDR-SB) score must be between 9.5 and 15.5.
3. Aged 55-80 years.
4. Must be receiving treatment with stable doses of acetylcholinesterase inhibitors, memantine, or both for at least 3 months prior to the screening visit.
5. Have a study partner who will provide written informed consent to participate, is in frequent contact with the participant (defined as at least 10 hours per week), and will accompany the participant to study visits or be available by telephone at designated times.
6. Have adequate literacy, vision, and hearing for neuropsychological testing in the opinion of the investigator at the time of screening.

Exclusion Criteria:

1. Has diagnosis of a clinically relevant central nervous system (CNS) disease other than AD dementia or other condition that negatively impacts cognition or cognitive status chronically.
2. Contraindications to MRI (e.g., metal implants) or inability to tolerate/comply with the scanning procedure.
3. Prior exposure to ozanimod or any other sphingosine-1-phosphate receptor regulators for AD before starting treatment with ozanimod subject of this study
4. Participants must not have clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, renal, infectious diseases, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult or that would put the participant at risk by participating in the study in the opinion of the Investigator.
5. Specific cardiac conditions are excluded, including history or presence of:

   i) Recent (within the past 6 months) occurrence of myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, New York Heart Association (NYHA) Class III/IV heart failure, or severe untreated sleep apnea.

   ii) Resting heart rate <55 beats per minute, second-degree (Mobitz type II) atrioventricular (AV) block, third-degree AV block, sick sinus syndrome, or sino-atrial block unless participants have a pacemaker in place.

   iii) Prolonged corrected QT interval by Fredericia's formula (QTcF; > 450 msec males and > 470 msec females), or participants at additional risk for QT prolongation.
6. Participants must not receive a live vaccine or a live-attenuated vaccine within 4 weeks prior to first dose or planning to receive a live vaccine or a live-attenuated vaccine during the study or within 90 days after discontinuation from study intervention.
7. Participants must not have a history of any significant drug allergy (such as anaphylaxis or hepatotoxicity).

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean Absolute Change From Baseline in Brain Amyloid Plaque on 18F-florbetaben PET Scan on Ozanimod Group Versus Control Group | Baseline to Week 27
  18F-florbetaben PET imaging was used as a quantitative amyloid biomarker. Quantitative amyloid burden was first formalized as the average Standardized Uptake Value Ratio (SUVR) in cortical areas of the brain relative to the cerebellum as a reference region. Larger SUVR reflects the larger cortical amyloid burden relative to cerebellum. SUVR values were further calibrated to a Centiloid (CL) scale. The Centiloid scale anchor points are 0 and 100, where 0 represents a high-certainty amyloid negative scan and 100 represents the amount of global amyloid deposition found in a typical AD scan. A negative change indicates an improvement from baseline.
Changes in serum GFAP | Baseline to Week 27
  We will quantify neuroinflammatory burden through plasma glial fibrillary acidic protein (GFAP) levels, comparing pre- and post-Ozanimod treatment, as well as between the Ozanimod group and the control group. Assessments will be conducted at baseline and week 27.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared due to the highly sensitive nature of genetic and biomarker profiles. De-identified aggregate data will be available upon reasonable request.